CLINICAL TRIAL: NCT07205835
Title: A Comparative Evaluation of the Effectiveness of an Artificial Intelligence-Generated Reformer Pilates Protocol and a Studio-Designed Reformer Pilates Protocol in Individuals With Forward Head Posture
Brief Title: Comparative Analysis of Artificial Intelligence-Generated and Studio-Based Reformer Pilates Interventions for Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Muhammed Fatih Kavak, Asst. Prof., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FZT2024/37
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Posture; Neck Disorder
Keywords: posture; Pain; Artificial intelligence (AI); Pilates exercises; Physiotherapy and rehabilitation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study population consisted of a total of 40 male and female volunteers aged between 18 and 50 years with a craniovertebral angle of less than 54 degrees. Participants were randomized into two groups: the Clinical Pilates group and the ChatGPT group. The Clinical Pilates group (n=20) performed clinical Pilates exercises under the supervision of a physiotherapist for 6 weeks, twice a week, 50 minutes per session. The ChatGPT group (n=20) followed an exercise program generated by ChatGPT under the supervision of a physiotherapist for 6 weeks, twice a week, 50 minutes per session.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Pilates Group (Experimental): Participants in this group will perform clinical Pilates exercises under the supervision of a physiotherapist, twice a week for 6 weeks. Each session will last 50 minutes and will include core stabilization, postural correction, and flexibility exercises.
  Interventions: Behavioral: Clinical Pilates Group
- ChatGPT Exercise Group (Active Comparator): Participants in this group will perform an exercise program generated by ChatGPT and supervised by a physiotherapist, twice a week for 6 weeks. Each session will last 50 minutes and will include exercises designed to improve posture, flexibility, and musculoskeletal function.
  Interventions: Behavioral: ChatGPT Exercise Group

INTERVENTIONS:
Behavioral: ChatGPT Exercise Group — Participants in the ChatGPT group will follow an exercise program generated by ChatGPT and supervised by a physiotherapist. The program will be delivered twice weekly for 6 weeks, with each 50-minute session including exercises designed to improve posture, flexibility, and musculoskeletal function.
  Arms: ChatGPT Exercise Group
Behavioral: Clinical Pilates Group — Participants in this arm will perform supervised clinical Pilates exercises twice weekly for 6 weeks. Each session will last 50 minutes and include core stabilization, postural correction, and flexibility exercises.
  Arms: Clinical Pilates Group

SUMMARY:
Posture is the alignment of body segments. While ideal posture places minimal stress on the joints, poor posture increases joint stress. Forward head posture (FHP) is a common postural abnormality characterized by the anterior displacement of the head in the sagittal plane. This condition may lead to muscle imbalances, pain, reduced cervical range of motion (ROM), decreased quality of life, and spinal degeneration.

The most common method for evaluating FHP is the craniovertebral angle (CVA). Causes of FHP include excessive smartphone and computer use, mouth breathing, carrying heavy bags, and rounded shoulders. Cervical stabilization exercises and holistic approaches are recommended for prevention and treatment.

Pilates, developed by Joseph Pilates, especially in its clinical form, has been shown to improve posture, strengthen core muscles, and enhance quality of life. Literature indicates that stretching- and strengthening-based exercise programs targeting FHP positively affect CVA, neck pain, and ROM.

In recent years, artificial intelligence (AI) has gained importance in physiotherapy as a diagnostic and therapeutic support tool. Its potential in generating exercise prescriptions is being explored, though whether AI can replace physiotherapists remains debated.

The aim of this study is to compare the effectiveness of an AI-generated reformer Pilates protocol and a studio-based reformer Pilates protocol in individuals with FHP. Hypotheses:

H0: The studio-based reformer Pilates protocol has no effect on CVA, ROM, pain, muscle endurance, or quality of life in individuals with FHP.

H1: The studio-based reformer Pilates protocol has a positive effect on these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Volunteers aged between 18-50 years

Craniovertebral angle less than 54°

Ability to participate in exercise sessions twice a week for 6 weeks

Willingness to provide informed consent

Exclusion Criteria:

History of musculoskeletal, neurological, or cardiovascular disorders

Previous surgery affecting posture or spine

Current participation in another structured exercise program

Pregnancy

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Change in Craniovertebral Angle | Baseline and after 6 weeks
  Craniovertebral angle will be measured using digital photography and goniometric analysis to evaluate postural improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Üsküdar Üniversitesi NP Sağlık Yerleşkesi, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. However, study results will be published in peer-reviewed scientific journals.